CLINICAL TRIAL: NCT04847219
Title: Efficacy and Safety of Premixed Insulin Treatment in Patients With Type 2 Diabetes Mellitus Observed by Different Type of Flash Glucose Mornitoring
Brief Title: Efficacy and Safety of Premixed Insulin Treatment in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Collaborators: Wuxi Hospital of Traditional Chinese Medicine (Unknown); Wuxi People's Hospital Affiliated to Nanjing Medical University (Unknown); Huai'an Second People's Hospital and the Affiliated Huai'an Hospital of Xuzhou Medical University (Unknown); The Affiliated Suqian First People's Hospital of Nanjing Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20190926-01
Record Dates: First submitted 2019-12-05; First posted 2021-04-19 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Professional flash glucose mornitoring (Placebo Comparator): Professional flash glucose mornitoring will be used in patients once a month for 3 months to monitor glucose level. Patients can learn their blood glucose levels via capillary blood glucose tests, but nor FGM duing FGM, and doctors will adjust their anti-diabetic therapy according to their FGM results after each monitoring.
  Interventions: Device: Professional flash glucose mornitoring
- Personal flash glucose mornitoring (Active Comparator): Personal flash glucose mornitoring will be used in patients once a month for 3 months to monitor glucose level. Patients can learn their blood glucose levels via FGM duing FGM, and doctors will adjust their anti-diabetic therapy according to their FGM results after each monitoring.
  Interventions: Device: Personal flash glucose mornitoring

INTERVENTIONS:
Device: Professional flash glucose mornitoring — Subjects will use Professional flash glucose mornitoring once a month for 3 months.
  Arms: Professional flash glucose mornitoring
Device: Personal flash glucose mornitoring — Subjects will use Personal flash glucose mornitoring once a month for 3 months.
  Arms: Personal flash glucose mornitoring

SUMMARY:
The aim of the study is to investigate the efficacy and safety of premixed insulin treatment in patients With type 2 diabetes mellitus using professional and personal Flash Glucose Mornitoring.

DETAILED DESCRIPTION:
Professional and personal Flash Glucose Mornitoring will be used in patients with type 2 diabetes who are treated with premixed insulin. The frequency of hypogycemia and the blood glucose control will be analyzed by flash glucose mornitoring once a month for 3 months and doctors will adjust the hypoglycemia treatment according to the results every month. HbA1c, glycemic variation, beta-cell function and androgen levels will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. participate voluntarily and sign the subject informed consent before the test.
2. for patients with type 2 diabetes who met WHO1999 diagnostic criteria, subcutaneous injection with premix insulin Bid/Tid, single drug and/or combination of oral hypoglycemic drugs, the treatment regimen was stable for more than 2 months.
3. no acute complications such as diabetic ketoacidosis and diabetic hyperosmolar syndrome.
4. subjects are able and willing to undergo FGM examination, diet and exercise regularly.

Exclusion Criteria:

1. patients treated with GLP-1 agonist in the last 3 months
2. patients who are allergic to insulin.
3. impaired liver and renal function, ALT 2.5 times higher than the upper limit of normal value;Serum creatinine was 1.3 times higher than the upper limit of normal.
4. a history of drug abuse and alcohol dependence within the past 5 years.
5. used systemic hormone therapy in recent 3 months.
6. patients with poor compliance and irregular diet and exercise.
7. patients with infection and stress within four weeks.
8. patients who cannot tolerate flash glucose mornitoring.
9. patients who are pregnant, nursing or or preparing to become pregnant.
10. any other apparent condition or comorption as determined by the investigator, such as severe heart and lung disease, endocrine disease, neurological disease, tumor disease, other pancreatic disease, history of mental illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
TIme in range | baseline and after 3 month
  change of TIme in range

SECONDARY OUTCOMES:
HbA1c | after 3 month
  change of glycated hemoglobin
antibody of insulin | baseline and after 3 month
  antibody of insulin
angrogen levels | baseline and after 3 month
  angrogen levels
exercise time daily | baseline and after 3 month
  duration of exercise daily
meal times | baseline and after 3 month
  daily times of meal
calorie intake | baseline and after 3 month
  daily calorie intake

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Ma, MD, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Kong D, Shen Z, Jiang L, Xie X, Yan R, Jing T, Hu Y, Ma J. The effects of vildagliptin on glycemic variability in patients with type 2 diabetes on premixed insulin therapy. Front Endocrinol (Lausanne). 2025 Jun 20;16:1508918. doi: 10.3389/fendo.2025.1508918. eCollection 2025. PMID 40620795
- [Derived] Yan RN, Cai TT, Jiang LL, Jing T, Cai L, Xie XJ, Su XF, Xu L, He K, Cheng L, Cheng C, Liu BL, Hu Y, Ma JH. Real-Time Flash Glucose Monitoring Had Better Effects on Daily Glycemic Control Compared With Retrospective Flash Glucose Monitoring in Patients With Type 2 Diabetes on Premix Insulin Therapy. Front Endocrinol (Lausanne). 2022 Feb 10;13:832102. doi: 10.3389/fendo.2022.832102. eCollection 2022. PMID 35222287
- [Derived] Cai T, Hu Y, Ding B, Yan R, Liu B, Cai L, Jing T, Jiang L, Xie X, Wang Y, Wang H, Zhou Y, He K, Xu L, Chen L, Cheng C, Ma J. Effect of Metformin on Testosterone Levels in Male Patients With Type 2 Diabetes Mellitus Treated With Insulin. Front Endocrinol (Lausanne). 2021 Dec 24;12:813067. doi: 10.3389/fendo.2021.813067. eCollection 2021. PMID 35002984